CLINICAL TRIAL: NCT07036198
Title: A User-Customizable Personalized Normative Feedback Intervention for Alcohol Harm Reduction in Young Adults: Feasibility, Acceptability, and Preliminary Efficacy
Brief Title: CPNF Intervention Development and Testing
Acronym: Project SHIFT
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Principal Investigator, Mary Larimer, Professor, University of Washington
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: STUDY00021161; R34AA031336 (NIH)
Record Dates: First submitted 2025-04-08; First posted 2025-06-25 (Actual); Last update posted 2025-07-17 (Actual); Status verified 2025-07

CONDITIONS: Alcohol Use
Keywords: young adults; alcohol-related harm; RCT; normative feedback
MeSH Terms: conditions — Alcohol Drinking

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- CPNF (Active Comparator): Customizable personalized normative feedback (CPNF) intervention whereby individuals can explore normative feedback for a wider variety of referent groups so that PNF is a truly personalized and engaging experience.
  Interventions: Behavioral: Customizable personalized normative feedback (CPNF)
- standard PNF (Active Comparator): Standard personalized normative feedback.
  Interventions: Behavioral: Personalized normative feedback (PNF)
- Attention-Matched Control (AMC) (Active Comparator): Attention-matched control.
  Interventions: Behavioral: Attention-Matched Control (AMC)

INTERVENTIONS:
Behavioral: Customizable personalized normative feedback (CPNF) — The CPNF intervention allows individuals to explore normative feedback for a wider variety of referent groups so that PNF is a truly personalized and engaging experience.
  Arms: CPNF
Behavioral: Personalized normative feedback (PNF) — Correcting misperceptions about peers' alcohol use behaviors and contrasting one's own use to the actual norms of their peers.
  Arms: standard PNF
Behavioral: Attention-Matched Control (AMC) — Participants in the AMC condition will complete all measures at the same time as participants in the CPNF condition but will not receive any information on drinking norms. Instead, participants in the AMC will receive normative feedback on sleep health, video game use, and gambling behaviors, and will similarly be able to choose the normative referent groups they wish to view feedback on for these behaviors. The AMC will thus serve as a non-treatment comparison that controls for assessment reactivity and effects of history and maturation.
  Arms: Attention-Matched Control (AMC)

SUMMARY:
The project will develop brief interventions that allow participants to customize which groups they receive feedback for in relation to things such as drinking norms for younger or older students, student athletes, etc. The goal is to provide content that is meaningful and engaging to all users.

DETAILED DESCRIPTION:
The project will develop and pilot test an innovative paradigm for leveraging social norms within brief interventions that entails user customization of which (and how many) normative referent groups they receive feedback for so that the content is meaningful and engaging to all users.

ELIGIBILITY:
Inclusion Criteria:

* Enrolled at the University of Washington either part- or full-time
* Report 3 or more past-month drinking occasions
* Report 3 or more drinks per occasion in the past month, on average
* Report 4 or more drinks during the peak drinking occasion in the past month
* Pass attention-check items

Exclusion Criteria:

N/A

Ages: 18 Years to 24 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 250 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2026-09-01 (Estimated); Study Completion 2027-09-01 (Estimated)

PRIMARY OUTCOMES:
Alcohol use - drinks per month | Screening, Baseline, Follow-ups, an average of 3 months
  Daily Drinking Questionnaire will assess drinks on average over the past month by recording the number of drinks consumed on each day of a typical week. Response options range from 0 drinks to 25+ drinks. Lower score is a better outcome, higher score is a worse outcome.
Alcohol use - Quantity per occasion | Screening, Baseline, Follow-ups, an average of 3 months
  Quantity/Frequency/Peak Alcohol Use Index will assess amount of alcohol consumed over the past month with how many days alcohol was consumed, average consumption, and peak consumption. Response options range from 0 to 30 days for frequency, and 1 to 12+ drinks for quantity and peak. Lower score is a better outcome, higher score is a worse outcome.
Alcohol use - Heavy episodic drinking | Screening, Baseline, Follow-ups, an average of 3 months
  Heavy Episodic Drinking measure will assess how many times over the past month heavy drinking episodes occurred, defined as 4 or more drinks (females) or 5 or more drinks (males) on a single occasion. Response options range from 0 to 7 days. Lower score is a better outcome, higher score is a worse outcome.
Alcohol use - Peak drinks & peak BAC | Screening, Baseline, Follow-ups, an average of 3 months
  Electronic Blood Alcohol content will be assessed and calculated using peak drinks over x amount of time. A lower BAC is a better outcome, a higher BAC is a worse outcome.
Alcohol use - Alcohol Use Disorders Identification Test | Baseline, Follow-ups, an average of 3 months
  The AUDIT is a 10-item self-report screening tool assessing hazardous and harmful alcohol use over the past year. Items are rated on varying 5-point Likert-type scales assessing frequency, quantity, and consequences of alcohol use. Lower score is a better outcome, higher score is a worse outcome.
Alcohol use - Brief Young Adult Alcohol Consequences Questionnaire | Baseline, Follow-ups, an average of 3 months
  The Brief YAACQ is a 24-item assessment of alcohol-related consequences in young adults. Response options for the items are yes or no. Higher score (i.e. more 'yes' responses) is a worse outcome, lower score (i.e. more 'no' responses) is a better outcome.

SECONDARY OUTCOMES:
Perceived descriptive norms for each normative referent group | Baseline, Follow-ups, an average of 3 months
  Gathered via Shortened Drinking Norms Rating Form. 7 items assess belief for what's an acceptable number of drinks each day of the week with responses ranging from 0 to 25+ drinks.
Perceived injunctive drinking norms for typical students at UW | Baseline, Follow-ups, an average of 3 months
  Gathered via the Injunctive Drinking Norms Rating Form. 7 items assess belief for what a typical UW college student drinks on each day of each day of the week with responses ranging from 0 to 25+ drinks.

CONTACTS AND LOCATIONS:
Overall Officials: Mary Larimer, PhD, Principal Investigator — University of Washington
Locations (1):
- The University of Washington, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: Yes
All scientific data (qualitative interview transcriptions, survey response data) will be both preserved and shared. Data will be made publicly available to the research community. This will include but may not be limited to (a) semi-structured interview questions, (b) survey items and corresponding response options (including missingness coding), (c) a codebook for scoring survey items and composite scales, (d) a detailed description of internally computed variables (e.g., time spent viewing intervention content), and (e) documentation of intervention components that participants were exposed to (both treatment and control conditions). Public use and restricted access study data and associated documentation will be made available to the research community free of charge through the NIAAA Data Archive.
Supporting Information: Study Protocol, ICF, Analytic Code
Time Frame: Data will be shared with the general research community at the time of an associated publication, or the end of the award/support period, whichever comes first.
Access Criteria: The data will be made available for sharing with the general research community via the NDA website. Investigators at institutions with a Federal Wide Assurance (FWA) will be able to gain access to NDA data by submitting a data access request in accordance with applicable NDA policies.